CLINICAL TRIAL: NCT04641494
Title: The Effect of 12 Weeks of Conjugated Linoleic Acid on Obesity Markers, Lung Functions, Lipid Profile and Inflammation in Overweight and Obese Women: Double-blind Randomised Control Trial.
Brief Title: The Effect of CLA on Obesity, Lung Functions, Lipid Profile and Inflammation in Women With BMI≥25
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1141/16/HH/CSN
Record Dates: First submitted 2020-09-16; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-08

CONDITIONS: Obesity; Lung Functions; Inflammation; Lipid Disorder
Keywords: Conjugated linoleic caid; Obesity; Lung functions; Inflammation; heat shock proteins; Adhesion molecules
MeSH Terms: conditions — Obesity; Inflammation; Lipid Metabolism Disorders | interventions — Linoleic Acids, Conjugated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): 28 subject received 2 capsules 3times a day for 12 weeks Each capsule contain 1gm (High Oleic Acid Safflower oils)
  Interventions: Dietary Supplement: High oleic acid safflower oil capsules
- CLA group (Active Comparator): Participants received 2 capsules3 times a day for 12 weeks Each capsule is 1 gm and it provided 0.75 gm CLA in a 50:50 mixture
  Interventions: Dietary Supplement: Conjugated linoleic acid

INTERVENTIONS:
Dietary Supplement: Conjugated linoleic acid — CLA Mixture capsule (50:50, c9, t11-CLA: t10, c12-CLA)
  Other Names: CLA
  Arms: CLA group
Dietary Supplement: High oleic acid safflower oil capsules
  Other Names: HOSFO
  Arms: Placebo

SUMMARY:
Conjugated linoleic acid or CLA, is one of the food supplements that could be found in meat, fats, and dairy products of ruminants which has been fed grass not on grains. CLA has shown anti-cancer, anti-obesity, and anti-inflammatory effects in several animal modules, but the results of the human studies were not consistent. Also, a very limited number of studies looked at the CLA effect on the respiratory system. The study will look at the effect of 12 weeks of supplementation of conjugated linoleic acid on obesity markers, lung functions, lipid profile, and inflammation in overweight and obese women in a double-blind randomized control trial.

The study looked at the inflammation using different approaches, where it looked at the expression of adhesion molecules on the proinflammatory monocytes as well as it analysed the expression of the stress proteins Heat-shock proteins (HSPA1A and HSPB1)on the PBMCs.

DETAILED DESCRIPTION:
This is a double-blind randomized control trial with parallel design, where consented overweight and obese women from Chester city in the UK will be randomly assigned into two groups one group CLA will receive 4.5 g/day CLA mixture capsules while the other group will receive a placebo.

Participants will attend three clinics and by the end of each clinic, the participants will be asked to provide 20 ml venous blood samples for the analysis of the biological marker. Participants' anthropometric, body composition, lung functions, Leptin adiponectin, lipid profile, Adhesion molecules CD14, CD16, CD11b, and CD62L, HSPA1A, and HSPB1 will be assessed at three time points, at baseline after 6 and 12 weeks. The level of CLA in the plasma, as well as lipid profile (HDL, LDL, TC, TG), will be measured at each time point

Participants will be asked to fill three food diaries before attending each clinic. Body composition will be measured using bioelectric impedance, lung functions will be assessed using spirometers, adiponectin and leptin will be assessed using ELISA, and finally, CD11b, CD62L, HSPA1A, and HSPB1 will be analysed using flow cytometer. Plasma level of c9, t11-CLA and t10, c12-CLA will be measured using flame ionized Gas chromatography, and the lipid profile will be assessed using ALERE AFINION™ AS100 ANALYZER.

Power calculation for the RCT Sample size calculation is done using G*Power software, a total of 20 participant is required, 10 participants in each group, to get an effect size of 1.3 kg/m2 change in BMI from baseline and SD of 0.45, 0.05 margin of error, 95% power and 95% confidence interval. Considering a 150% drop out the total number will be 50, 25 in each group.

Participants' randomisation will be performed by an independent third party who is not involved in the current trial. Participants will be randomised into blocks using (www.randomization.com) which generate the randomisation plan. All the capsules will be packed in a light protective dark brown tamper-proof container. The randomised participants will be either allocated to the CLA group or the placebo group. CLA and placebo capsules will have the same shape and colour, and both the participants and researcher will be blind to the treatments.

Statistical analysis. IBM SPSS Statistic Data Editor Software (version25) will be used for the statistical analysis of this trial while the graphs will be made using GraphPad Prism version 7.

Descriptive statistics of baseline continuous data will be expressed in form of mean± standard error of the mean (SEM). Nominal data will be expressed in percentages. The parametric assumption will be checked using Shapiro-Wilk tests at a significant level p< 0.05. The differences between the baseline characteristics in CLA and the placebo group will be done using an independent t-test in parametric data or Mann Whitney U for non-parametric data, at a significant level P<0.05.

Testing the effects of CLA compared to placebo and the interaction with times (baseline, 6 weeks, and 12 weeks) will be done using Mixed Model Repeated Measures Analysis of Variance (ANOVA) at a significant level p< 0.05. The later analysis will be useing Tukey post hoc test with Bonferroni correction for all the measured parameters.

A paired t-test or Wilcoxon test will be done to detect the difference within- participants at different time points in parametric and non-parametric data, respectively, at a significant level P<0.05. Independent t-test or Mann Whitney U will be used to detect the difference between the CLA group and placebo across the different time points for normally and non-normally distributed data, respectively at a significant level P<0.05.

The difference in the change at week 6 compared to baseline, (∆ 6 weeks), and at week 12 compared to baseline (∆ 12 weeks), in CLA groups compared to placebo will be checked using t-test in case of normally distributed data or Mann Whitney-U for non-parametric data at significant level P<0.05. The difference between the categorical data will be done using the Chi-square test at a significant level p<0.05.

Obesity hypotheses

H1: There is a significant reduction in BMI in CLA supplemented group compared to the placebo group.

H0: There is no significant reduction in BMI in CLA supplemented group compared to the placebo group.

H2: There is a significant reduction in BW in the CLA supplemented group compared to the placebo group.

H0: There is no significant reduction in BW in the CLA supplemented group compared to the placebo group.

H3: There is a significant reduction in WHR in CLA supplemented group compared to the placebo group.

H0: There is no significant reduction in WHR in CLA supplemented group compared to the placebo group.

H5: There is a significant increase in LBM in CLA supplemented group compared to the placebo group.

H0: There is no significant increase in LBM in CLA supplemented group compared to the placebo group.

H6: There is a significant increase in %LBM in CLA supplemented group compared to the placebo group.

H0: There is no significant increase in %LBM in CLA supplemented group compared to the placebo group.

H8: There is a significant reduction in TBF in CLA supplemented group compared to the placebo group.

H0: There is no significant reduction in TBF in CLA supplemented group compared to the placebo group.

H9: There is a significant reduction in %BF in CLA supplemented group compared to the placebo group.

H0: There is no significant reduction in %BF in CLA supplemented group compared to the placebo group.

H10: There is a significant increase in the basal metabolic rate in the CLA supplemented group compared to the placebo group.

H0: There is no significant increase in the basal metabolic rate in the CLA supplemented group compared to the placebo group.

Lung function hypotheses Primary hypothesis H1: There is a significant increase in %PEF predicted in CLA supplemented group compared to the placebo group.

H0: There is no significant increase in %PEF predicted in CLA supplemented group compared to the placebo group.

Secondary hypotheses. H2: There is a significant increase in %FEV1 predicted in CLA supplemented group compared to the placebo group.

H0: There is no significant increase in %FEV1 predicted in CLA supplemented group compared to the placebo group.

H3: There is a significant increase in %FVC predicted in CLA supplemented group compared to the placebo group.

H0: There is no significant increase in %FVC predicted in CLA supplemented group compared to the placebo group.

H8: There is a significant increase in %FEV1/FVC predicted in CLA supplemented group compared to the placebo group.

H0: There is no significant increase in %FEV1/ FVC predicted in CLA supplemented group compared to the placebo group.

8.6.3 Adipokines hypotheses Primary hypothesis H1: There is a significant reduction in leptin in the CLA supplemented group compared to the placebo group.

H0: There is no significant reduction in leptin in the CLA supplemented group compared to the placebo group.

Secondary hypothesis. H2: There is a significant increase in adiponectin in the CLA supplemented group compared to the placebo group.

H0: There is no significant increase in adiponectin in the CLA supplemented group compared to the placebo group.

8.6.4 Inflammation hypotheses Primary hypothesis H1: there is a significant change in the expression of HSPA1A on PBMCs in the CLA group compared to the placebo group.

H0: there is no significant change in the expression of HSPA1A on PBMCs in the CLA group compared to the placebo group.

Secondary hypotheses H2: there is a significant change in the expression of HSPA1A on lymphocytes in the CLA group compared to the placebo group.

H0: there is no significant change in the expression of HSPA1A on lymphocytes in the CLA group compared to the placebo group.

H3: there is a significant change in the expression of HSPA1A on monocytes in the CLA group compared to the placebo group.

H0: there is no significant change in the expression of HSPA1A on monocytes in the CLA group compared to the placebo group.

H4: there is a significant change in the expression of HSPB1on PBMCs in the CLA group compared to the placebo group.

H0: there is no significant change in the expression of HSPB1 on PBMCs in the CLA group compared to the placebo group.

H5: there is a significant change in the expression of HSPB1 on lymphocytes in the CLA group compared to the placebo group.

H0: there is no significant change in the expression of HSPB1 on lymphocytes in the CLA group compared to the placebo group.

H6: there is a significant change in the expression of HSPB1 on monocytes in the CLA group compared to the placebo group.

H0: there is no significant change in the expression of HSPB1 on monocytes in the CLA group compared to the placebo group.

H7: there is a significant change in the expression of CD11b on pro-inflammatory monocytes (CD14++CD16+) in the CLA group compared to the placebo group.

H0: there is no significant change in the expression of CD11b on pro-inflammatory monocytes (CD14++CD16+) in the CLA group compared to the placebo group.

H8: there is a significant change in the expression of CD11b on pro-inflammatory monocytes (CD14++CD16+) after 100ng/ml LPS stimulation for one hour in the CLA group compared to the placebo group.

H0: there is no significant change in the expression of CD11b on pro-inflammatory monocytes (CD14++CD16+) in the CLA group compared to the placebo group.

H9: there is a significant change in the increase of CD11b expression on pro-inflammatory monocytes (CD14++CD16+) after LPS stimulation in the CLA group compared to the placebo group.

H0: there is no significant difference H8: there is a significant change in the increase of CD11b expression on pro-inflammatory monocytes (CD14++CD16+) after LPS stimulation in the CLA group compared to the placebo group.

H10: there is a significant change in the expression of CD62L on pro-inflammatory monocytes (CD14++CD16+) in the CLA group compared to the placebo group.

H0: there is no significant change in the expression of CD62L CD11b on pro-inflammatory monocytes (CD14++CD16+) in the CLA group compared to the placebo group.

H11: there is a significant change in the expression of CD62L on pro-inflammatory monocytes (CD14++CD16+) after 100ng/ml LPS stimulation for one hour in the CLA group compared to the placebo group.

H0: there is no significant change in the expression of CD62L on pro-inflammatory monocytes (CD14++CD16+) in the CLA group compared to the placebo group.

H12: there is a significant change in the reduction of CD62L expression on pro-inflammatory monocytes (CD14++CD16+) after LPS stimulation in the CLA group compared to the placebo group.

H0: there is no significant change in the reduction of CD62L expression on pro-inflammatory monocytes (CD14++CD16+) after LPS stimulation in the CLA group compared to the placebo group.

Lipid profile hypotheses H1: there is a significant change in the level of LDL in the CLA group compared to the placebo group.

H0: there is no significant change in the level of LDL in the CLA group compared to the placebo group.

H2: there is a significant change in the level of HDL in the CLA group compared to the placebo group.

H0: there is no significant change in the level of HDL in the CLA group compared to the placebo group.

H3: there is a significant change in the level of TC in the CLA group compared to the placebo group.

H0: there is no significant change in the level of TC in the CLA group compared to the placebo group.

H4: there is a significant change in the level of TG in the CLA group compared to the placebo group.

H0: there is no significant change in the level of TG in the CLA group compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Able to swallow capsules
* Overweight and obese women (BMI≥25)
* Forced expiratory volume FEV1≥ 70%

Exclusion Criteria:

* Participants taking antibiotics,
* Participants taking weight loss medications
* Pregnant and breastfeeding women,
* Women with current or a history of severe lung disease

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
The change in body weight from baseline to 12 weeks | 0, 6, 12 Weeks
  Body weight (Kg) will be measured using Bioelectric impedance technique (Tanita MC-780)
The change in BMI from baseline to 12 weeks | 0, 6, 12 Weeks
  weight and height will be combined to report BMI in kg/m^2
The change in total body fat from baseline to 12 weeks | 0, 6, 12 Weeks
  total body fat (Kg) will be measured using Bioelectric impedance technique (Tanita MC-780)
The change in percentage body fat from baseline to 12 weeks | 0, 6, 12 Weeks
  Percentage body fat will be measured using Bioelectric impedance technique (Tanita MC-780)
The change in Lean body mass from baseline to 12 weeks | 0, 6, 12 Weeks
  Lean body mass (Kg) will be measured using Bioelectric impedance technique (Tanita MC-780)
The change in percentage lean body mass from baseline to 12 weeks | 0, 6, 12 Weeks
  Percentage lean body mass will be measured using Bioelectric impedance technique (Tanita MC-780)
The change in waist circumference from baseline to 12 weeks | 0, 6, 12 Weeks
  Waist circumference will be measured by cm using the tab
The change in waist to hip ratio from baseline to 12 weeks | 0, 6, 12 Weeks
  Waist to hip ratio will be calculated by dividing the waist circumference cm over the hip circumference

SECONDARY OUTCOMES:
The change in Total Cholesterol (TC) from baseline to 12 weeks | 0, 6, 12 weeks
  TC mmol/l was measured by (Alere Afinion™ AS100 Analyzer)with test cartridges (Alere Afinion™ Lipid Panel).
The change in Triglycerides (TG) from baseline to 12 weeks | 0, 6, 12 weeks
  TG (mmol/l)was measured by (Alere Afinion™ AS100 Analyzer)with test cartridges (Alere Afinion™ Lipid Panel).
The change in Low Density Lipoprotein (LDL) from baseline to 12 weeks | 0, 6, 12 weeks
  LDL (mmol/l) was measured by (Alere Afinion™ AS100 Analyzer)with test cartridges (Alere Afinion™ Lipid Panel).
The change in (High Density Lipoprotein) HDL from baseline to 12 weeks | 0, 6, 12 weeks
  HDL (mmol/l) was measured by (Alere Afinion™ AS100 Analyzer) with test cartridges (Alere Afinion™ Lipid Panel).

OTHER OUTCOMES:
The change in (Forced Expiratory Volume) FEV% predicted from baseline to 12 weeks | 0, 6, 12 weeks
  was measured using Micro loop spirometer
The change in (Forced Vital Capacity) FVC% predicted from baseline to 12 weeks | 0, 6, 12 weeks
  was measured using Micro loop spirometer
The change in (Peak of Flow) PEF% predicted from baseline to 12 weeks | 0, 6, 12 weeks
  was measured using Micro loop spirometer
The change in expression of CD11b on pro-inflammatory monocytes (CD14++CD16+) from baseline to 12 weeks | 0, 6, 12 weeks
  CD11b (MFI) expression was measured using Flow cytometer
The change in expression of CD62L on pro-inflammatory monocytes (CD14++CD16+) from baseline to 12 weeks | 0, 6, 12 weeks
  CD62L (MFI) expression was measured using Flow cytometer
The change in the plasma level of Leptin from baseline to 12 weeks | 0,6,12 weeks
  Leptin (ng/ml) was measured using commercially available ELISA
The change in the plasma level of Adiponectin from baseline to 12 weeks | 0,6,12 weeks
  Adiponectin (µg/ml) was measured using commercially available ELISA
The change in expression of HSPA1A on PBMCs from baseline to 12 weeks | 0, 6, 12weeks
  HSPA1A (MFI) expression was measured using Flow cytometer
The change in expression of HSPB1 on PBMCs from baseline to 12 weeks | 0, 6, 12weeks
  HSPB1 (MFI) expression was measured using Flow cytometer
The change in plasma level of c9,t10-CLA from baseline to 12 weeks | 0, 6, 12 weeks
  C9,t11-CLA (µg/ml) level will be measured using flam ionised gas chromatography
The change in plasma level of t10, c12-CLA from baseline to 12 weeks | 0, 6, 12 weeks
  T10, c12-CLA (µg/ml) level will be measured using flam ionised gas chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Hanady Hamdallah, PhD, Principal Investigator — University of Chester
Locations (1):
- University of Chester, Chester, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The results will be available in the thesis form and possibly publication. It will be available in the thesis form in 2022 and publication expected to be in 2021.